CLINICAL TRIAL: NCT06194994
Title: Emotion Regulation as a Moderator of Two Different Treatments for Children With Oppositional Defiant Disorder: A Randomized Clinical Trial
Brief Title: Emotion Regulation as a Moderator of Two Different Treatments for Children With ODD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Urdur Njardvik, Professor, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UI-2023-ODDEMREG
Record Dates: First submitted 2023-06-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Oppositional Defiant Disorder
Keywords: Oppositional Defiant Disorder; Emotion Regulation; Child Psychopathology
MeSH Terms: conditions — Oppositional Defiant Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomisation to two different treatments which will be compared.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers and outcomes assessors will be blind to emotion regulation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Training (Experimental): Behavioral parent training intervention. Individual sessions.
  Interventions: Behavioral: Parent Management Training
- Child directed treatment (Experimental): Child directed cognitive behavioral therapy. Individual sessions.
  Interventions: Behavioral: Tuning Your Temper

INTERVENTIONS:
Behavioral: Parent Management Training — Behavioral parent training program aimed at increasing compliance and positive behaviours while decreasing disruptive behaviours
  Arms: Parent Training
Behavioral: Tuning Your Temper — Cognitive behavioural treatment for children focusing on arousal reduction, problem solving and cognitive restructuring.
  Arms: Child directed treatment

SUMMARY:
The goal of this randomized controlled trial is to is to test emotion regulation as a moderator of two different treatments for children with Oppositional Defiant Disorder (ODD). The main question it aims to answer is whether treatment gains be increased when children with ODD receive a treatment congruent with their emotion regulation skill problems. Participants will be divided into two groups based on their response patterns; a high emotion dysregulation group and a low emotion dysregulation group. Within each group, children will then be randomly assigned to either a behavioral parent training intervention or a child directed treatment involving problem solving and emotion regulation skills.

DETAILED DESCRIPTION:
Emotion regulation has been implicated in the development of ODD. Two types of treatment are commonly used for children with ODD, behavioral parent training and child directed cognitive treatments. Parent training focuses on increasing compliance and reducing defiant behaviour while the child directed treatments focus on increasing the child's problem solving skills and emotion regulation. The investigators will assess emotion regulation and emotional lability in children diagnosed with ODD and divide them into two groups based on their response patterns; a high emotion dysregulation group and a low emotion dysregulation group. Within each group, children will then be randomly assigned to either a behavioral parent training intervention or a child directed treatment involving problem solving and emotion regulation skills, which makes it possible to assess the effects of the different interventions for the two distinct groups. Treatment effects will be assessed at pre- and post-treatment as well as at 6 and 18 month follow-up. Comorbid conditions will be tested as moderators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Oppositional Defiant Disorder
* Icelandic speaking (child and parent/guardian)

Exclusion Criteria:

* IQ below 70 (full scale score)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Disruptive Behaviour Rating Scale | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Parent and teacher rated questionnaire to assess change in symptoms of ODD.
Schedule for Affective Disorders and Schizophrenia for School Aged Children (K-SADS-PL) | Pre-treatment; 6-month follow-up; 18-month follow-up.
  Diagnostic Interview to assess whether a child changes in diagnostic status, whether child meets DSM-5 diagnostic criteria for mental disorders.

SECONDARY OUTCOMES:
Strength and difficulties questionnaire | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Parent and teacher rated questionnaire to assess change in emotional and behavioral problems. Results are converted to t-scores where t=65 is considered a clinical cut-off score. Higher scores indicate worse outcome.
Home Situations Questionnaire | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Parent rated questionnaire to assess change in compliance and problematic behaviour at home. Frequency of problems is recorded (min 0, max 16) and severity score for each item endorsed is rated on the scale of 0-9 with higher scores indicating worse outcome.
Social Skills Rating System | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Parent rated questionnaire to assess change in social skills. The SSRS has 55 questions rated from 0-2 (min 0 max 110). There are 4 social skills domains: Cooperation, Assertion, Responsibility and Self-control with higher scores indicating better outcome. And 3 problem domains (External, Internal and Hyperactivity) with higher scores indicating worse outcome.
Parent Stress Index | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Parent rated questionnaire to assess change in parental stress. Scores range from 18-90 with higher scores indicating higher levels of parental stress.
Pediatric Quality of Life Index | Pre-treatment; Immediately post-treatment; 6-month follow-up; 18-month follow-up.
  Questionnaire to assess change in child quality of life. The parent version used has 23 items rated on a scale from 0-4 (min 0 max 92). High scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Urdur Njardvik, PhD, Principal Investigator — Department of Psychology, University of Iceland
Locations (1):
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No
As the study includes repeated measures of a vulnerable population, parts of the data will be classified as sensitive personal data and thus restricted by the permit from the Bioethics Committee. We will consult with GAGNÍS (member of CESSDA ERIC) on how to make the data available according to the FAIR principles.

REFERENCES:
- [Background] Njardvik U, Smaradottir H, Ost LG. The Effects of Emotion Regulation Treatment on Disruptive Behavior Problems in Children: A Randomized Controlled Trial. Res Child Adolesc Psychopathol. 2022 Jul;50(7):895-905. doi: 10.1007/s10802-022-00903-7. Epub 2022 Feb 8. PMID 35133557
- [Background] Barkley, R. A. (2013). Defiant children: A clinician's manual for assessment and parent training: Guilford press